CLINICAL TRIAL: NCT00453544
Title: Enhancing Consent for Alzheimer's Research
Acronym: BWP-AD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Barton W. Palmer, Ph.D., Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IA0110; 1R01AG028827 (NIH)
Record Dates: First submitted 2007-03-28; First posted 2007-03-29 (Estimated); Results first posted 2023-06-06 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Alzheimer Disease
Keywords: computer assisted instruction; decision making; educational resource design /development; executive function
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Enhanced consent - A (Experimental): The intervention was an enhanced consent process, including a multimedia aid for a moderate risk hypothetical protocol
  Interventions: Other: Enhanced Consent Procedure
- Enhanced consent - B (Experimental): The intervention was an enhanced consent process, including multimedia aide for a higher risk hypothetical protocol
  Interventions: Other: Enhanced Consent Procedure
- Routine consent - A (Active Comparator): This was a comparison condition - a routine consent process, including a printed consent document, for a moderate risk hypothetical protocol
  Interventions: Other: Routine Consent Procedure
- Routine consent - B (Active Comparator): This was a comparison condition - a routine consent process, including a printed consent document, for a higher risk hypothetical protocol
  Interventions: Other: Routine Consent Procedure

INTERVENTIONS:
Other: Enhanced Consent Procedure — This is a procedure involving use of multimedia materials, as well as standard review with research staff, to see if the research consent procedure can be improved
  Arms: Enhanced consent - A; Enhanced consent - B
Other: Routine Consent Procedure — This is a procedure designed to be in accord with standard research consent practices (and lacks multimedia aids)
  Arms: Routine consent - A; Routine consent - B

SUMMARY:
The purpose of this study is to evaluate the efficacy of an enhanced consent procedure for patients with mild-to-moderate Alzheimer disease, and to identify factors and patient characteristics that predict the degree to which enhanced consent is more beneficial than routine consent procedures.

DETAILED DESCRIPTION:
Alzheimer disease can impair the capacity of patients to give informed consent for research participation. Studies of informed consent involving other patient populations suggest better understanding of consent-relevant information may be achieved through modifications in the consent delivery process, including incorporation of multimedia learning tools into the consent discussion.

In the present study, participants with Alzheimer disease and age-comparable healthy participants will be randomly assigned to review a hypothetical research protocol via routine or enhanced consent procedures. Participants will also complete standard cognitive and other rating scales so that we can characterize the sample, as well as evaluate the degree to which specific characteristics may be associated with need for enhanced consent procedures. Advances in the methods to optimize the informed consent process should enable future research participants to make more fully informed decisions.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of mild to moderate possible or probable AD or demographically comparable healthy comparison subjects
* Fluency in English
* 50 yrs and older
* Informed written consent (or written assent with consent from legally authorized representative)

Exclusion Criteria:

* Diagnosis of Lewy Body Dementia or Mild Cognitive Impairment
* MMSE less than 15
* Physical or medical conditions that preclude participants from completing tasks
* Healthy comparison volunteers if they have a known neurologic or psychiatric condition that could impair neurocognitive functioning

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2006-04; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barton W. Palmer, PhD, Principal Investigator — UCSD
Locations (1):
- Veterans Affairs San Diego Healthcare System, San Diego, California, United States

REFERENCES:
- [Background] Kim SY, Caine ED, Currier GW, Leibovici A, Ryan JM. Assessing the competence of persons with Alzheimer's disease in providing informed consent for participation in research. Am J Psychiatry. 2001 May;158(5):712-7. doi: 10.1176/appi.ajp.158.5.712. PMID 11329391
- [Background] Alzheimer's Association. Research consent for cognitively impaired adults: recommendations for institutional review boards and investigators. Alzheimer Dis Assoc Disord. 2004 Jul-Sep;18(3):171-5. doi: 10.1097/01.wad.0000137520.23370.56. PMID 15494623
- [Background] Kolata G. Alzheimer's research poses dilemma. Science. 1982 Jan 1;215(4528):47-8. doi: 10.1126/science.7053558.
- [Background] Dunn LB, Jeste DV. Enhancing informed consent for research and treatment. Neuropsychopharmacology. 2001 Jun;24(6):595-607. doi: 10.1016/S0893-133X(00)00218-9. PMID 11331139
- [Result] Palmer BW, Harmell AL, Pinto LL, Dunn LB, Kim SY, Golshan S, Jeste DV. Determinants of Capacity to Consent to Research on Alzheimer's disease. Clin Gerontol. 2017;40(1):24-34. doi: 10.1080/07317115.2016.1197352. Epub 2016 Jun 7. PMID 28154452
- [Result] Palmer BW, Harmell AL, Dunn LB, Kim SY, Pinto LL, Golshan S, Jeste DV. Multimedia Aided Consent for Alzheimer's Disease Research. Clin Gerontol. 2018 Jan-Feb;41(1):20-32. doi: 10.1080/07317115.2017.1373177. Epub 2017 Nov 28. PMID 29182458

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Enhanced Consent - A | Enhanced Consent - B | Routine Consent - A | Routine Consent - B
Started | 62 | 55 | 68 | 67
Completed | 60 | 54 | 68 | 66
Not Completed | 2 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Not completed — Primary outcome measure not completed | 1 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: 259 subjects met inclusion/exclusion criteria, but 8 withdrew prior to the randomization (only two due to study - i.e. 2 found assessments too frustrating); 3 additional subjects had missing data key outcomes; resulting in 248 subjects in the final data analysis..
Groups:
- Total: Total of all reporting groups
Arm/Group | Enhanced Consent - A | Enhanced Consent - B | Routine Consent - A | Routine Consent - B | Total
Number analyzed (Participants) | 60 | 54 | 68 | 66 | 248
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 3 | 6 | 7 | 20
  >=65 years | 56 | 51 | 62 | 59 | 228
Age, Continuous [Mean (Standard Deviation); unit: years] | 78.4 (8.5) | 79.5 (8.4) | 79.3 (8.3) | 78.4 (8.5) | 78.9 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 25 | 31 | 35 | 124
  Male | 27 | 29 | 37 | 31 | 124
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 0 | 2 | 1 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 2 | 4 | 10
  White | 56 | 49 | 63 | 58 | 226
  More than one race | 1 | 0 | 2 | 1 | 4
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants] — All participants were recruited and seen in the San Diego, CA metropolitan area.
  participants
    United States | 60 | 54 | 68 | 66 | 248

OUTCOME MEASURES:

1. Primary Outcome: Level of Understanding
Description: Modified version of the MacArthur Competence Assessment Tool for Clinical Research (MacCAT-CR) Understanding subscale.
  Minimum value = 0, Maximum value = 26; higher scores represent better performance
Time Frame: Within session - administered approximately 2-3 minutes after completion of the simulated consent process.
Population: 114 people with Alzheimer's disease (AD); 134 non-neuropsychiatric comparison (NC) subjects; the effects of routine vs. enhanced consent and moderate vs. higher risk were analyzed within diagnostic groups separately
Measure: Mean (Standard Deviation); unit: score on a scale (MacCAT-CR Und Trial 2)
Groups:
- AD Enhanced Consent - Mod Risk: Group = participants with mild-to-moderate AD
  The intervention was an enhanced consent process, including a multimedia aid for a moderate risk hypothetical protocol
  Enhanced Consent Procedure: This is a procedure involving use of multimedia materials, as well as standard review with research staff, to see if the research consent procedure can be improved
- AD Enhanced Consent - Higher Risk: Group = participants with mild-to-moderate AD
  The intervention was an enhanced consent process, including multimedia aide for a higher risk hypothetical protocol
  Enhanced Consent Procedure: This is a procedure involving use of multimedia materials, as well as standard review with research staff, to see if the research consent procedure can be improved
- AD Routine Consent - Mod Risk: Group = participants with mild-to-moderate AD
  This was a comparison condition - a routine consent process, including a printed consent document, for a moderate risk hypothetical protocol
  Routine Consent Procedure: This is a procedure designed to be in accord with standard research consent practices (and lacks multimedia aids)
- AD Routine Consent - Higher Risk: Group = participants with mild-to-moderate AD
  This was a comparison condition - a routine consent process, including a printed consent document, for a higher risk hypothetical protocol
  Routine Consent Procedure: This is a procedure designed to be in accord with standard research consent practices (and lacks multimedia aids)
- NC Enhanced Consent - Mod Risk: Group = NC subjects
  The intervention was an enhanced consent process, including a multimedia aid for a moderate risk hypothetical protocol
  Enhanced Consent Procedure: This is a procedure involving use of multimedia materials, as well as standard review with research staff, to see if the research consent procedure can be improved
- NC Enhanced Consent - Higher Risk: Group = NC subjects
  The intervention was an enhanced consent process, including multimedia aide for a higher risk hypothetical protocol
  Enhanced Consent Procedure: This is a procedure involving use of multimedia materials, as well as standard review with research staff, to see if the research consent procedure can be improved
- NC Routine Consent - Mod Risk: Group = NC subjects
  This was a comparison condition - a routine consent process, including a printed consent document, for a moderate risk hypothetical protocol
  Routine Consent Procedure: This is a procedure designed to be in accord with standard research consent practices (and lacks multimedia aids)
- NC Routine Consent - Higher Risk: Group = NC subjects
  This was a comparison condition - a routine consent process, including a printed consent document, for a higher risk hypothetical protocol
  Routine Consent Procedure: This is a procedure designed to be in accord with standard research consent practices (and lacks multimedia aids)
Arm/Group | AD Enhanced Consent - Mod Risk | AD Enhanced Consent - Higher Risk | AD Routine Consent - Mod Risk | AD Routine Consent - Higher Risk | NC Enhanced Consent - Mod Risk | NC Enhanced Consent - Higher Risk | NC Routine Consent - Mod Risk | NC Routine Consent - Higher Risk
Number analyzed (Participants) | 26 | 24 | 33 | 31 | 34 | 30 | 35 | 35
score on a scale (MacCAT-CR Und Trial 2) | 17.8 (7.0) | 16.8 (7.6) | 15.1 (6.9) | 15.7 (7.7) | 25.2 (1.1) | 24.8 (2.2) | 25.3 (1.1) | 24.9 (2.3)

2. Primary Outcome: Appreciation
Description: MacArthur Competence Assessment Tool for Clinical Research (MacCAT-CR) Appreciation subscale Minimum score = 0, Maximum Score = 6; Higher scores represent better understanding
Time Frame: Within session - immediately following administration of the MacCAT-CR Understanding subscale
Population: 114 people with Alzheimer's disease (AD); 132 non-neuropsychiatric comparison (NC) subjects; the effects of routine vs. enhanced consent and moderate vs. higher risk were analyzed within diagnostic groups separately
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AD Enhanced Consent - Mod Risk | AD Enhanced Consent - Higher Risk | AD Routine Consent - Mod Risk | AD Routine Consent - Higher Risk | NC Enhanced Consent - Mod Risk | NC Enhanced Consent - Higher Risk | NC Routine Consent - Mod Risk | NC Routine Consent - Higher Risk
Number analyzed (Participants) | 26 | 24 | 33 | 31 | 33 | 30 | 35 | 34
score on a scale | 4.2 (1.8) | 4.2 (1.6) | 4.2 (1.3) | 4.1 (1.7) | 5.5 (0.8) | 4.7 (1.1) | 5.2 (1.0) | 5.1 (1.1)

3. Primary Outcome: Reasoning
Description: Reasoning subscale of the MacArthur Competence Assessment Tool for Clinical Research (MacCAT-CR) Minimum score = 0; Maximum Score = 8; Higher scores mean better reasoning capacity
Time Frame: Within session-immediately following administration of the MacCAT-CR Appreciation subscale
Population: 112 people with Alzheimer's disease (AD); 133 non-neuropsychiatric comparison (NC) subjects; the effects of routine vs. enhanced consent and moderate vs. higher risk were analyzed within diagnostic groups separately
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- AD Enhanced Consent - Mod Risk: Group = participants with mild-to-moderate Alzheimer's Disease (AD)
  The intervention was an enhanced consent process, including a multimedia aid for a moderate risk hypothetical protocol
  Enhanced Consent Procedure: This is a procedure involving use of multimedia materials, as well as standard review with research staff, to see if the research consent procedure can be improved
- AD Enhanced Consent - Higher Risk: Group = participants with mild-to-moderate Alzheimer's Disease (AD)
  The intervention was an enhanced consent process, including multimedia aide for a higher risk hypothetical protocol
  Enhanced Consent Procedure: This is a procedure involving use of multimedia materials, as well as standard review with research staff, to see if the research consent procedure can be improved
- AD Routine Consent - Mod Risk: Group = participants with mild-to-moderate Alzheimer's Disease (AD)
  This was a comparison condition - a routine consent process, including a printed consent document, for a moderate risk hypothetical protocol
  Routine Consent Procedure: This is a procedure designed to be in accord with standard research consent practices (and lacked multimedia aids)
- AD Routine Consent - Higher Risk: Group = participants with mild-to-moderate Alzheimer's Disease (AD)
  This was a comparison condition - a routine consent process, including a printed consent document, for a higher risk hypothetical protocol
  Routine Consent Procedure: This is a procedure designed to be in accord with standard research consent practices (and lacks multimedia aids)
- NC Enhanced Consent - Mod Risk: Group = non-neuropsychiatric comparison (NC) subjects
  The intervention was an enhanced consent process, including a multimedia aid for a moderate risk hypothetical protocol
  Enhanced Consent Procedure: This is a procedure involving use of multimedia materials, as well as standard review with research staff, to see if the research consent procedure can be improved
- NC Enhanced Consent - Higher Risk: Group = non-neuropsychiatric comparison (NC) subjects
  The intervention was an enhanced consent process, including multimedia aide for a higher risk hypothetical protocol
  Enhanced Consent Procedure: This is a procedure involving use of multimedia materials, as well as standard review with research staff, to see if the research consent procedure can be improved
- NC Routine Consent - Mod Risk: Group = non-neuropsychiatric comparison (NC) subjects
  This was a comparison condition - a routine consent process, including a printed consent document, for a moderate risk hypothetical protocol
  Routine Consent Procedure: This is a procedure designed to be in accord with standard research consent practices (and lacks multimedia aids)
- NC Routine Consent - Higher Risk: Group = non-neuropsychiatric comparison (NC) subjects
  This was a comparison condition - a routine consent process, including a printed consent document, for a higher risk hypothetical protocol
  Routine Consent Procedure: This is a procedure designed to be in accord with standard research consent practices (and lacks multimedia aids)
Arm/Group | AD Enhanced Consent - Mod Risk | AD Enhanced Consent - Higher Risk | AD Routine Consent - Mod Risk | AD Routine Consent - Higher Risk | NC Enhanced Consent - Mod Risk | NC Enhanced Consent - Higher Risk | NC Routine Consent - Mod Risk | NC Routine Consent - Higher Risk
Number analyzed (Participants) | 26 | 23 | 33 | 30 | 34 | 30 | 35 | 34
score on a scale | 6.9 (1.5) | 6.2 (2.5) | 5.6 (2.5) | 6.3 (2.4) | 7.6 (0.7) | 7.5 (0.8) | 7.3 (1.3) | 7.5 (0.9)

4. Primary Outcome: Expression of a Choice
Description: Expression of a Choice subscale of the MacArthur Competence Assessment Tool for Clinical Research (MacCAT-CR); Minimum score = 0, Maximum score = 2; higher scores represent more intact ability to express a clear choice
Time Frame: Within session--immediately following administration of the MacCAT-CR Reasoning subscale
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AD Enhanced Consent - Mod Risk | AD Enhanced Consent - Higher Risk | AD Routine Consent - Mod Risk | AD Routine Consent - Higher Risk | NC Enhanced Consent - Mod Risk | NC Enhanced Consent - Higher Risk | NC Routine Consent - Mod Risk | NC Routine Consent - Higher Risk
Number analyzed (Participants) | 26 | 23 | 33 | 30 | 34 | 30 | 35 | 34
units on a scale | 1.8 (0.6) | 1.7 (0.7) | 1.7 (0.6) | 1.5 (0.8) | 1.9 (0.2) | 2.0 (0.0) | 1.9 (0.2) | 1.9 (0.3)

5. Secondary Outcome: Level of Satisfaction With Consent Process
Description: Question - "The consent process was" rated from "Very easy" to "Very Hard"
  1. Very Easy
  2. Easy
  3. No effect
  4. Hard
  5. Very hard Higher scores mean more difficult (less satisfaction) with the consent process
     * with 1 being "Very Easy" and 5 being "Very hard"
Time Frame: Within session
Population: Administered immediately after the MacCAT-CR Expression of a Choice subscale
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AD Enhanced Consent - Mod Risk | AD Enhanced Consent - Higher Risk | AD Routine Consent - Mod Risk | AD Routine Consent - Higher Risk | NC Enhanced Consent - Mod Risk | NC Enhanced Consent - Higher Risk | NC Routine Consent - Mod Risk | NC Routine Consent - Higher Risk
Number analyzed (Participants) | 20 | 15 | 24 | 21 | 33 | 30 | 34 | 32
score on a scale | 1.3 (2.1) | 2.4 (1.9) | 2.0 (2.1) | 1.9 (2.1) | 1.9 (0.9) | 1.8 (0.6) | 1.7 (0.6) | 1.7 (0.6)

6. Secondary Outcome: Expressed Willingness to Participate in the Hypothetical Protocol
Description: Question about willingness to consent in the protocol described 0 = No
  1. = Yes
  2. = Unsure
Time Frame: Within session-last item of the Expression of a Choice Subscale, which itself was measured immediately after the MacCAT-CR Reasoning subscale
Population: 111 people with Alzheimer's disease (AD); 131 non-neuropsychiatric comparison (NC) subjects; the effects of routine vs. enhanced consent and moderate vs. higher risk were analyzed within diagnostic groups separately
Measure: Number; unit: percentage of yes
Arm/Group | AD Enhanced Consent - Mod Risk | AD Enhanced Consent - Higher Risk | AD Routine Consent - Mod Risk | AD Routine Consent - Higher Risk | NC Enhanced Consent - Mod Risk | NC Enhanced Consent - Higher Risk | NC Routine Consent - Mod Risk | NC Routine Consent - Higher Risk
Number analyzed (Participants) | 25 | 24 | 31 | 31 | 33 | 30 | 35 | 33
percentage of yes | 76 | 83 | 81 | 71 | 79 | 67 | 54 | 56

ADVERSE EVENTS:
Time Frame: Adverse Events were not monitored/assessed.
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | Enhanced Consent - A | Enhanced Consent - B | Routine Consent - A | Routine Consent - B
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No